CLINICAL TRIAL: NCT03805087
Title: Transarterial Coil Embolization of the Superior Rectal Arteries for Treatment of Stage II Hemorrhoids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICH-Emborrhoid
Record Dates: First submitted 2018-12-24; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Hemorrhoids; Embolization, Therapeutic
Keywords: Hemorrhoids; Embolization, Therapeutic
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coil embolization (Experimental): Transarterial coil embolization of the superior rectal arteries via a transradial left arterial access.
  Interventions: Procedure: Transarterial coil embolization

INTERVENTIONS:
Procedure: Transarterial coil embolization — Transarterial coil embolization of the superior rectal arteries via a transradial left arterial access.

SUMMARY:
This study will evaluate short , mid and long term efficacy of transarterial coil embolization of the superior rectal arteries (Emborrhoid techinque) for treatment the hemorrhoidal disease.

DETAILED DESCRIPTION:
The 'emborrhoid' technique is the embolization of the hemorrhoidal arteries. The endovascular arterial occlusion is performed using coils placed in the terminal branches of the superior rectal arteries The emborrhoid technique has been modeled after elective transanal Doppler-guided hemorrhoidal artery ligation, which has been shown to be safe and effective for hemorrhoidal disease.

To date, there are few reports regarding emborrhoid, particularly lacking in long-term follow-up. Additionally, all procedures reported so far have used a transfemoral access route, which requires at least one day of hospital stay.

The aims of this study are:

To increase data regarding safety and efficacy of the Emborrhoid technique To report changes in the quality of life of patients at short and long-term To quantify recurrences at one-year follow-up To validate the use of the radial access for the Emborrhoid technique To validate the Emborrhoid technique as a "one-day" hospital procedure

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least grade II Hemorrhoids (Banov et al. 1985), agreeing to undergo the Embhorroid technique.

Exclusion Criteria:

* Absolute contraindications to an angiographic procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the severity of symptoms of hemorrhoidal disease | 1 years
  A symptom-based severity score (Sordegren scoring system) will be used before and after intervention. It is a questionnaire composed by 4 questions with a final scoring of 0-14 where 14 is the highest possible severity of symptoms.
  The questionnaire will be administered the day before procedure, one week after procedure and one year after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: EZIO LANZA, MD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Humanitas Research Hospital, Rozzano, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Berczi V, Gopalan D, Cleveland TJ. Embolization of a hemorrhoid following 18 hours of life-threatening bleeding. Cardiovasc Intervent Radiol. 2008 Jan-Feb;31(1):183-5. doi: 10.1007/s00270-006-0179-4. PMID 17334848
- [Result] Vidal V, Louis G, Bartoli JM, Sielezneff I. Embolization of the hemorrhoidal arteries (the emborrhoid technique): a new concept and challenge for interventional radiology. Diagn Interv Imaging. 2014 Mar;95(3):307-15. doi: 10.1016/j.diii.2014.01.016. Epub 2014 Feb 28. PMID 24589187
- [Result] Tradi F, Louis G, Giorgi R, Mege D, Bartoli JM, Sielezneff I, Vidal V. Embolization of the Superior Rectal Arteries for Hemorrhoidal Disease: Prospective Results in 25 Patients. J Vasc Interv Radiol. 2018 Jun;29(6):884-892.e1. doi: 10.1016/j.jvir.2018.01.778. Epub 2018 Apr 30. PMID 29724519